CLINICAL TRIAL: NCT02733640
Title: Does Pantoprazole Reduce the Anti-platelet Effect of Clopidogrel?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, PI (professor), Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B-1112/141-006
Record Dates: First submitted 2016-03-28; First posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Antiplatelet Effect
MeSH Terms: interventions — Pantoprazole; Ranitidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Pantoprazole (Active Comparator): Drug: Pantoprazole 40 mg once-daily
  Interventions: Drug: Pantoprazole
- Ranitidine (Experimental): Drug: Ranitidine 150 mg twice-daily
  Interventions: Drug: Ranitidine

INTERVENTIONS:
Drug: Pantoprazole — pantoprazole 40 mg once-daily
  Arms: Pantoprazole
Drug: Ranitidine — ranitidine 150 mg twice-daily
  Arms: Ranitidine

SUMMARY:
The investigators sought to evaluate the influence of pantoprazole, indicated as less effective than other proton pump inhibitors, on the antiplatelet effect of clopidogrel, with stratification of the population according to the presence of cytochrome (CYP) 2C19 polymorphism.

DETAILED DESCRIPTION:
Participants being treated with a maintenance dose of 75 mg clopidogrel and 100 mg aspirin daily after previous PCI with coronary stenting were included in the study. Participants were randomly assigned to either the pantoprazole 40 mg once-daily group or the ranitidine 150 mg twice-daily group using a computer-generated randomized table. An independent investigator generated the random allocation sequence. Blood samples were collected at 9:00 on day prior to treatment (day 0) and on day 9. Measuring impedance was performed by one independent investigator in a blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated with a maintenance dose of 75 mg clopidogrel and 100 mg aspirin daily after previous PCI with coronary stenting were included in the study. All patients received standardized therapy with a loading dose of 600 mg of clopidogrel hydrogen sulfate and 400 mg aspirin.

All participants had a normal platelet count (150,000-450,000/mL).

Exclusion Criteria:

* Patients with severe liver disorders, current gastrointestinal disorders, a current infection, congestive heart failure, or a known bleeding disorder as well as patients on bivalirudin or glycoprotein IIb/III antagonists within the last 7 days were excluded from the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with more than 5 Ω of impedance after intervention by an aggregometer which measures platelet aggregation in whole blood samples | 8 days
  8 days after administration of pantoprazole (or ranitidine)

SECONDARY OUTCOMES:
Change of the impedance value (Ω) by an aggregometer which measures platelet aggregation in whole blood samples | baseline and 8days
  8 days after administration of pantoprazole (or ranitidine)
Number of participants with gastrointestinal bleeding | up to 2weeks
Number of participants with reccured coronary artery disease | up to 2weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Choi YJ, Kim N, Jang IJ, Cho JY, Nam RH, Park JH, Jo HJ, Yoon H, Shin CM, Park YS, Lee DH, Jung HC. Pantoprazole Does Not Reduce the Antiplatelet Effect of Clopidogrel: A Randomized Controlled Trial in Korea. Gut Liver. 2017 Jul 15;11(4):504-511. doi: 10.5009/gnl16352. PMID 28395507